CLINICAL TRIAL: NCT04977609
Title: Music in Action: A Music-based Virtual Reality Intervention for Upper Limb Motor Rehabilitation in Post-stroke Hemiparetic Patients
Brief Title: A Music-based VR Intervention for Upper Limb Motor Rehabilitation in Hemiparetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione Poliambulanza (Unknown)
Responsible Party: Principal Investigator, Alice Cancer, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUSIC-IN-ACTION
Record Dates: First submitted 2021-07-03; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Hemiparesis
Keywords: Music; Motor coordination; Embodied cognition; Rehabilitation; Virtual reality; Action observation
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR+MUSIC (Experimental): Upper limb repetitive training activities through the imitation of movements (i.e., unscrew the cap of a bottle, pour water into a glass, drink water from a glass, sugaring coffee, placing an object in a box) synchronized with a musical accompaniment (i.e., a selection of classical music pieces). Participants will wear a VR headset (Gear VR, Samsung) through which they will observe egocentric 180° 3D videoclips shot from a first-person perspective, as if the patient himself was performing the movement, while listening to music.
  Interventions: Behavioral: VR+MUSIC
- VR (Experimental): Upper limb repetitive training activities through imitation of movements, without any musical accompaniment. Participants will wear a VR headset through which they will observe egocentric 180° 3D silent videoclips.
  Interventions: Behavioral: VR
- TAU (Active Comparator): Treatment as usual (TAU). Patients will be engaged in upper limb repetitive training activities through traditional physiotherapy rehabilitation.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: VR+MUSIC — A novel VR intervention designed for upper limb motor rehabilitation in post-stroke hemiparetic patients consisting in 10 daily sessions of 30 minutes, over 2 weeks, supervised by a physical therapist.
  Arms: VR+MUSIC
Behavioral: VR — A novel VR intervention designed for upper limb motor rehabilitation in post-stroke hemiparetic patients consisting in 10 daily sessions of 30 minutes, over 2 weeks, supervised by a physical therapist.
  Arms: VR
Behavioral: TAU — Traditional post-stroke upper limb motor rehabilitation under the supervision of a physical therapist, for 0 daily sessions of 30 minutes, over 2 weeks.
  Arms: TAU

SUMMARY:
Hemiparesis affects the majority of stroke patients in the acute phase. In post-stroke motor rehabilitation patients can re-learn motor sequences through repetitive training. Research showed that virtual reality (VR) can be effectively used in upper limb motor rehabilitation by training motor coordination and gestures in an immersive virtual environment. Another promising line of intervention in post-stroke rehabilitation is the use of music, with evidence supporting the notion that a rhythmic accompaniment promotes the recovery of motor coordination in patients with hemiparetic stroke. Furthermore, studies showed a beneficial effect of the observation of movements performed by a third person in patients with post-stroke hemiparesis. Based this evidence, the present study aims at testing the feasibility and efficacy of a novel music-based VR intervention designed for upper limb motor rehabilitation in post-stroke hemiparetic patients. The treatment consists in upper limb repetitive training activities through the imitation of movements synchronized with a musical accompaniment and is delivered in 10 sessions over 2 weeks, supervised by a physical therapist. Participants wear a VR headset through which they observe egocentric 180° 3D videoclips. The experimental condition (group A) will be compared with a no-music condition (group B), to test the specific effect of music, and with traditional physiotherapy rehabilitation (group C), to test the efficacy of the approach. The investigators expect that the patients undergoing the experimental intervention (group A and group B) will show a greater upper limb motor function improvement, as compared to the active control group. As a secondary endpoint the investigators expect the music component to induce a greater motor improvement as compared to the experimental condition without music.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke patients in acute/subacute phase
* Upper limb hemiparesis (Ashworth scale: 0-2; MRC scale: 3-5)
* Age between 18 and 80 years
* Currently enrolled in inpatient rehabilitation

Exclusion Criteria:

* Psychiatric disorders,
* Neglect
* Epilepsy
* MMSE rating < 24
* Difficulty with visual-spatial exploration
* Visual deficits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Motricity Index (Collin, 1990) | 2 weeks post-test
  Motricity scale
Medical Research Council (MRC) Muscle strength scale (Paternostro-Slug et al., 2008) | 2 weeks post-test
  Muscle strenght scale
The Chedoke arm and Hand Activity Inventory (CAHAI) - short form (Barreca, 2013) | 2 weeks post-test
  Hand activity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Poliambulanza, Brescia, Italy